CLINICAL TRIAL: NCT02660528
Title: Tocilizumab Augmentation in Treatment-Refractory Major Depressive Disorder: An Open-Label Trial
Brief Title: Tocilizumab Augmentation in Treatment-Refractory Major Depressive Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study staff change.
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jessica Harder, Associate Psychiatrist, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015P001263
Record Dates: First submitted 2016-01-19; First posted 2016-01-21 (Estimated); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tocilizumab (Experimental): Tocilizumab 162 mg sc q2weeks x 4 doses
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Subcutaneous tocilizumab
  Other Names: Actemra

SUMMARY:
This proposed study sets out to examine the antidepressant effects of tocilizumab among patients with treatment-refractory major depression.

DETAILED DESCRIPTION:
As the understanding of the complex relationship between pro-inflammatory cytokines (specifically interleukin-6 [IL-6]) and depression symptoms becomes clearer, clinical trials to evaluate effective and novel treatments are needed. As there have been no published tocilizumab trials among patients with major depression, this pilot study will adopt a single-arm, open-label design. Due to the notion that inflammatory cytokines may play a role in a sub-type of depression, this study will recruit patients with treatment refractory major depressive disorder, for whom established depression treatments have not been effective. In conducting this trial, the investigators seek to examine the potential role of tocilizumab as an augmentation agent, with the hypothesis that it could reduce depression symptomatology in patients with major depression who have not experienced symptom reduction through more traditional antidepressant therapies.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of major depressive episode
* Hamilton Depression Rating Scale (HDRS) score of >20
* In treatment for depression for a minimum of 8 weeks

Exclusion criteria:

* Active drug or alcohol disorder in the last three months
* History of psychosis, mania or hypomania
* Acute suicide or homicide risk
* History of liver disease including HCV and HBV
* HIV
* History of heart disease or a heart attack
* Active or latent tuberculosis, a history of a positive tuberculosis test, or having received the Bacillus Calmette-Guérin (BCG) vaccine
* Epilepsy or a history of seizures
* Abnormal thyroid-stimulating hormone (TSH <0.4 or >5.0mlU/L)
* Abnormal liver function tests on screening (ALT>50 U/L or AST>50 U/L)
* Low absolute neutrophil count (ANC) on screening (<4000/mm3
* Abnormal white blood cell count (<4,500 or > 10,000mcL)
* Low platelet count on screening (<150,000/mm3
* Patients with an active or recent infection, for example cellulitis, bacteremia, pneumonia, and pyelonephritis.
* Recent exposure to uncommon infections (e.g. histoplasmosis, blastomycosis, coccidiomycosis) through recent travel to the Ohio and Mississippi River Valleys and the Southwest
* Pregnant women, breastfeeding women or women of child-bearing age not using contraception
* History of or current autoimmune disease, including multiple sclerosis and inflammatory bowel disease
* Diagnosis of chronic fatigue syndrome
* Temperature greater than 100.3F at the screening visit or any subsequent visits
* Dyslipidemia
* Currently taking oral steroids
* Currently taking statins
* Chronic aspirin or NSAID takers
* Currently taking any immunomodulating medications
* Inability to consent due to cognitive impairment

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Harder, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Sukoff Rizzo SJ, Neal SJ, Hughes ZA, Beyna M, Rosenzweig-Lipson S, Moss SJ, Brandon NJ. Evidence for sustained elevation of IL-6 in the CNS as a key contributor of depressive-like phenotypes. Transl Psychiatry. 2012 Dec 4;2(12):e199. doi: 10.1038/tp.2012.120. PMID 23212583
- [Background] Al-Hakeim HK, Al-Rammahi DA, Al-Dujaili AH. IL-6, IL-18, sIL-2R, and TNFalpha proinflammatory markers in depression and schizophrenia patients who are free of overt inflammation. J Affect Disord. 2015 Aug 15;182:106-14. doi: 10.1016/j.jad.2015.04.044. Epub 2015 May 5. PMID 25985379
- [Background] Fonseka TM, McIntyre RS, Soczynska JK, Kennedy SH. Novel investigational drugs targeting IL-6 signaling for the treatment of depression. Expert Opin Investig Drugs. 2015 Apr;24(4):459-75. doi: 10.1517/13543784.2014.998334. Epub 2015 Jan 14. PMID 25585966

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were assigned to treatment arms because none of the participants were eligible to continue the study after screening.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Baseline Demographics: Demographics of screened subjects.
Arm/Group | Baseline Demographics
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.67 (2.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change on Hamilton Depression Rating Scale (HDRS)
Description: Absolute change on Hamilton Depression Rating Scale (HDRS) score
Time Frame: Baseline to 8 Weeks
Population: No data was collected for the study outcome measures because none of the participants were eligible to continue the study after screening.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 0

2. Secondary Outcome: Proportion of Subjects Achieving Remission (HDRS Score < 7)
Description: Proportion of Subjects with an HDRS score < 7
Time Frame: 8 Weeks
Population: as for outcome 1
Arm/Group | Tocilizumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Proportion of Subjects Achieving Response (HDRS Score Decreased >50% From Baseline)
Description: Proportion of Subjects with an HDRS score decreased >50% from baseline
Time Frame: 8 Weeks
Population: as for outcome 1
Arm/Group | Tocilizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were not collected as no participants were eligible to participate in the study after screening.
Description: No adverse event information was recorded because no participants were eligible to continue with the study after screening.
Arm/Group | Tocilizumab
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT02660528/Prot_SAP_000.pdf